CLINICAL TRIAL: NCT03829163
Title: Efficacy and Cost Effectiveness of Utilizing a Hydraulically Adjustable Walker in the Treatment of Hip Fracture
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB -- need to reframe study as a feasibility study before it being a RCT.
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Peter Klausmeyer, Principal Investigator, MaineHealth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: klausmeyerHAW
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: This study is a randomized prospective, parallel, voluntary study to test the effectiveness of a newly designed stair-climbing walker on post-acute care patients with hip fractures. Consecutive patients participating in the study will be given participant numbers 1- 40 (odd numbered participant numbers = conventional walker, even numbered participant numbers = HAW) to protect their privacy and to eliminate selection bias. They each will receive training on each assistive device via their assigned inpatient physical therapist. The HAW should not be kept in a vehicle overnight or in temperatures below 45 degrees due to possible hydraulic system failures. A standard walker will be offered along with the HAW to the even numbered patients to ensure that the patient will have an assistive device after the study is completed or if there was an issue with the HAW during the study and needed to be discontinued.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Walker Group (Active Comparator)
  Interventions: Device: Conventional Walker
- HAW Group (Experimental)
  Interventions: Device: Hydraulic Adjustable Walker

INTERVENTIONS:
Device: Hydraulic Adjustable Walker — The HAW is a based on a conventional walker but has innovative telescoping legs with a leg adjustment assembly that includes at least one valve and at least one tube that delivers hydraulic fluid into the legs and allows a user to control the length of each leg. The legs of the walker are hydraulically adjustable, so that the front legs may be shortened and the back legs extended, or two side legs shortened and the two opposing side legs extended, so as to allow the walker to be securely placed on two different steps. This allows the user to be able to stand on a stair without worrying about sharing the same stair with the device. It also ensures that the height of the walker continues to be the right height for the user to minimize loss of balance.
  Arms: HAW Group
Device: Conventional Walker — A walker consists primarily of a metal frame with four legs which are stabilized by crossbars. These walker frames come in a variety of shapes and sizes; many consist primarily of two inverted U-shaped leg modules connected by crossbars. Regardless of the shape or form of the leg modules, each walker frame forms a 3-sided box with an opening in which the user may stand.
  Arms: Conventional Walker Group

SUMMARY:
The purpose of this study is to establish the efficacy of a new walker with hydraulically adjustable legs (HAW) in increasing patients' mobility, especially over uneven terrains such as stairs. An attempt will be made to determine patients' satisfaction with this new instrument as well as comparing it to current walkers' effects on mobility, patient confidence, safety and security. In addition, an estimate of financial advantages/savings will be reviewed. Patient using the HAW should benefit from increased mobility, increased freedom home and in the community, as well as decreased medical costs and need for home modifications along with burden on family members caring for them after the injury.

DETAILED DESCRIPTION:
Assistive walking devices are well known and come in various forms, such as canes, crutches, and walkers. Their primary purpose has been to allow someone to be more functional, safe, and independent after a sudden or gradual decline in some aspect of their health. Even with vast changes in all areas of human development the standard walking devices still have their limitations especially when it comes to stairs. The HAW takes one of the most common and dependable devices, a conventional walker, and upgrades its functionality to handle stairs and uneven ground.

A walker consists primarily of a metal frame with four legs which are stabilized by crossbars. These walker frames come in a variety of shapes and sizes; many consist primarily of two inverted U-shaped leg modules connected by crossbars. Regardless of the shape or form of the leg modules, each walker frame forms a 3-sided box with an opening in which the user may stand (See Figure 1).

The frame often includes two handles located on each side of the user at the upper region of each inverted U-shaped member. The height is matched to each individual's height by keeping the handles at the height of their inner wrist (See Figure 1).

Most basic walkers include mechanical means to allow the length of the legs to be increased or decreased. Push button locking pins that fit into pre-drilled holes in the legs are used to secure the walkers height to match the person [HO10] using it. The adjustment is also a time-consuming process requiring significant dexterity, and if a patient is trying to do it themselves, this can lead to falls or injury.

The US spends over $30 billion on health care-related to falls each year. 1 There are over 1,000,000 hip and knee surgeries performed each year. 1 In the US, the National Institute of Health (NIH) estimates that there are 6.9 million assistive device users (crutches, canes, or walker) in the US patient that are over the age of 65. 1 Currently there is an estimated 2 million walker users. It is estimated that of those 2 million, 62% of them have to use a walker to navigate stairs on a daily basis.1 This means that conservatively 1.24 million elderly people would benefit from a walker that negotiates stairs optimally. This number of elderly people will undoubtedly be increasing as the elderly population is estimated to more than double by the year 2050, reaching an astounding 89,000,000. 1 The HAW is the only known device that would allow its user the safety of a standard walker as well as protection on stairs while maintaining or improving their muscle strength, balance and endurance. 1 The HAW is a based on a conventional walker but has innovative telescoping legs with a leg adjustment assembly that includes at least one valve and at least one tube that delivers hydraulic fluid into the legs and allows a user to control the length of each leg. The legs of the walker are hydraulically adjustable, so that the front legs may be shortened and the back legs extended, or two side legs shortened and the two opposing side legs extended, so as to allow the walker to be securely placed on two different steps. This allows the user to be able to stand on a stair without worrying about sharing the same stair with the device. It also ensures that the height of the walker continues to be the right height for the user to minimize loss of balance.

The design has been tested to be able to withstand 300 pounds of force per leg without failure, so a conservative maximum load would be 600 lbs. Hydraulics were used instead of a mechanical designed to allow for infinite number of adjustments for varying stair heights. A standard stair is 8.25 inches tall, but can range from 6 inches up to 9 inches in some homes. The HAW allows for a wide variety of stairs to be able to be fit with a single adjustment instead of the multiple adjustments required with a conventional walker or crutch.

Dwaine Philbrook, PT, and Director of Rehab for Coastal Health Care Alliance of Maine, commented on the HAW: "In 32 years of clinical practice this is one of the most innovative medical products that I have ever seen. The biggest obstacle for patients returning home from a hospital stay, that require a walker, is how to negotiate stairs. Many are unable to use crutches due to balance issues or general weakness. The hydraulic walker will enable those patients to safely use stairs and enjoy a higher level of functional mobility" (May, 2016 personal communication to author).

It is anticipated that the study should confirm that patients using the HAW on stairs and for general mobility should improve the patient's satisfaction after the initial injury, improve their fear of falling again, and give them the confidence and ability to become an active member in their community earlier than those with a convention walker. Daily logs completed by the patients should show improved ambulation distances as compared to the control group which will improve the patients recovery and decrease need for further healthcare costs.

The use of the HAW for patients with an acute hip fracture should improve the patient's recovery and possibly decrease time spent in the hospital following the injury. The HAW will reduce the need for costly home repairs while improving a patient's fear of falling on stairs, improve their community ambulation, decrease medical bills, and lower the need for assistance from outside people within the home.

Using data that is collected by the study coordinator from the patient themselves, and their scores on the functional outcome measures in the tables below, the studies aim is to show an accelerated recovery and return to a prior level of function faster than the control group. This data along with the patient's testimonials will hopefully show that the HAW can be used for a wide variety of patients to improve their level of mobility and safety during ambulation on stairs along with uneven ground.

Conventional walkers are not well suited or functionally intended for use on stairways or uneven surfaces. The inability of conventional walkers to allow patients to properly balance on such surfaces limits their usefulness and may introduce significant risk to the user. There exists a need for a walker that allows its user to have safety, stability, control, and ease of use for navigating inclined, declined or uneven surfaces. Thus, the Hydraulically Adjustable Stair Climbing Walker (HAW) was developed.

ELIGIBILITY:
Inclusion Criteria:

* 1. 40 consecutive mentally competent patients (as determined by a score of 22 or higher on the mini mental state exam.) 2. Patients age 65-90 who suffer an acute hip fracture from a fall and will be assigned to the use of a walker. The patient will be given and instructed on the use of the Waldo County General Hospital standard walker or the HAW.

Exclusion Criteria:

* 1. Patients who are deemed cognitively impaired (scores less than 22 on mini mental state exam).

  2. Patients who are unable to lift a walker up onto steps. 3. Patients who have upper extremity weakness or injury due to fall and unsafe to use a standard walker as intended.

  4. Patient who are shorter than five foot two inches tall or patients six foot three inches or taller as height limitations are based on prototypes available at this time.

Early withdrawal can be done at any time by a patient for any reason especially if the patient feels unsafe with the assigned walker or if surgery is indicated for a non-union of the fracture or failure of the implanted TFN.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with improved balance using the HAW assessed by Berg Balance Scale | 24 months
  Berg Balance Scale About: This scale measures balance in older adults. Items: 14
  Equipment:
  Yardstick One standard chair with arm rests One standard chair without arm rests Footstool/step Stopwatch or wristwatch 15 foot walkway Reliability: Cronbach's alphas were greater than 0.83 for stroke patients and 0.97 for elderly residents.
  Scoring:
  A five-point scale, a range of 0-4. 0 = lowest level of function 4 = highest level of function. Highest possible score = 56 Score of < 45 indicates a greater risk of falling 41-56 = low fall risk 21-40 = medium fall risk 0 -20 = high fall risk
  Reference:
  Berg K, Wood-Dauphinee S, Williams JI, Maki, B (1992). Measuring balance in the elderly: validation of an instrument. Can. J. Pub. Health July/August supplement 2:S7-11
  Norms:
  Lusardi, M.M. (2004). Functional Performance in Community Living Older Adults. Journal of Geriatric Physical Therapy, 26(3), 14-22.
Number of Participants with improved mobility using the HAW assessed by Lower Extremity Functional Scale | 24 months
  The Lower Extremity Functional scale (LFES) is a self-administered set of 20 questions with answers ranging from 0-4 to assess the function of one or both lower extremities. The rating scale is as follows:
  0. Extreme difficulty, including inability to perform an activity
  1. Quite a bit of difficulty
  2. Moderate difficulty
  3. A little bit of difficulty
  4. No difficulty The totals are summed at the bottom of the table. The minimum important change on the scale is 9 points, which means that a clinical change exists with a change of 9 points on the scale.
  The LEFS has a margin of error of +/- 5 points, which means that a patient's tabulated score is within 5 points of his "true" score.
Number of participants with accelerated recovery | 24 Months
  Using data that is collected by the study coordinator from patients involved in the study, and their scores on the functional outcome measures in the tables below, the study aim is to show an accelerated recovery and return to a prior level of function among use of the HAW faster than the control group using a conventional walker. This data, along with patient testimonials, will hopefully show that the HAW can be used for a wide variety of patients to improve their level of mobility and safety during ambulation on stairs and uneven ground.

SECONDARY OUTCOMES:
Number of participants with reduced costs associated with the HAW | 24 Months
  The HAW will reduce the need for costly home repairs, while improving a patient's fear of falling on stairs, improve their community ambulation, decrease medical bills, and lower the need for assistance from outside people within the home.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klausmeyer, PT, DPT, Principal Investigator — Waldo County General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] University of California - Disability Statistics Center. (2018, September 28). Mobility Device Statistics: United States. Retrieved October 3, 2018, from https://www.disabled-world.com/disability/statistics/mobility-stats.php
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- See also: Official Website for the "HAW" -- invited and built by one of the investigators of 3 Wills, LLC. — https://3willswalkers.wixsite.com/walker